CLINICAL TRIAL: NCT03709121
Title: An Exploratory Clinical Trial Evaluating Reproxalap Ophthalmic Solutions (0.25% and 0.5%) in Subjects With Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC)
Brief Title: A Methodology Development Clinical Trial of Reproxalap in Subjects With Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-011
Record Dates: First submitted 2018-10-03; First posted 2018-10-17 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-10

CONDITIONS: Conjunctivitis, Allergic
Keywords: reproxalap; ADX-102; allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Reproxalap Ophthalmic Solution (0.5%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.5%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) dosed twice.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Reproxalap Ophthalmic Solution (0.5%) — Reproxalap Ophthalmic Solution (0.5%) dosed twice.
  Arms: Reproxalap Ophthalmic Solution (0.5%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution dosed twice.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
An Exploratory Clinical Trial Evaluating Reproxalap Ophthalmic Solutions (0.25% and 0.5%) in Subjects with Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC)

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race
* have at least a two-year history of moderate-to-severe ragweed-induced allergic conjunctivitis based on principal investigator's judgement
* have a positive skin prick test to ragweed pollen within the past year of screening

Exclusion Criteria:

* known contraindication or hypersensitivities to any components of the investigational product medication or components
* history of uveitis, blepharitis, dry eye syndrome, herpes simplex keratitis, or herpes zoster keratitis;
* presence of any ocular infection (bacterial, viral, or fungal) or active ocular inflammation (e.g., follicular conjunctivitis, allergic conjunctivitis) within 14 days prior to screening
* presence of any chronic ocular degenerative condition or ocular inflammation that, in the opinion of the investigator, is likely to worsen over the course of the clinical trial;
* presence of any chronic ocular degenerative condition or ocular inflammation that, in the opinion of the investigator, is likely to worsen over the course of the clinical trial
* diagnosis of moderate-to-severe pinguecula or pterygium (particularly if it results in chronic erythema), Stevens-Johnson Syndrome, ocular cicatricial pemphigoid, mucous membrane pemphigoid, significant conjunctival scarring, chemical burn, herpetic or neurotrophic keratitis, Cryopyrin Associated Periodic Syndrome (CAPS), or keratoconus
* woman of childbearing potential who is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inflamax Research Limited, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy subjects were randomized in a three-way crossover design trial.
Groups:
- Reproxalap (0.25%), Then Reproxalap (0.5%), Then Vehicle: Reproxalap (0.25%) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day washout (Washout #1), then Reproxalap (0.5%) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day (Washout #2), then Vehicle was administered once 5 minutes before and 90 minutes after allergen chamber entry.
- Reproxalap (0.5%), Then Vehicle, Then Reproxalap (0.25%): Reproxalap (0.5%) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day washout (Washout #1), then Vehicle was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day (Washout #2), then Reproxalap (0.25%) was administered once 5 minutes before and 90 minutes after allergen chamber entry.
- Vehicle, Then Reproxalap (0.25%), Then Reproxalap (0.5%): Vehicle was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day washout (Washout #1), then Reproxalap (0.25%) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day (Washout #2), then Reproxalap (0.5%) was administered once 5 minutes before and 90 minutes after allergen chamber entry.
Period: Overall Study
Arm/Group | Reproxalap (0.25%), Then Reproxalap (0.5%), Then Vehicle | Reproxalap (0.5%), Then Vehicle, Then Reproxalap (0.25%) | Vehicle, Then Reproxalap (0.25%), Then Reproxalap (0.5%)
Started | 22 | 25 | 23
Completed | 22 | 22 | 22
Not Completed | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Reproxalap (0.5%), Then Vehicle, Then Reproxalap (0.25%): Reproxalap (0.5%) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day washout (Washout #1), then Vehicle) was administered once 5 minutes before and 90 minutes after allergen chamber entry, then there was a 14-day (Washout #2), then Reproxalap (0.25%) was administered once 5 minutes before and 90 minutes after allergen chamber entry.
- Total: Total of all reporting groups
Arm/Group | Reproxalap (0.25%), Then Reproxalap (0.5%), Then Vehicle | Reproxalap (0.5%), Then Vehicle, Then Reproxalap (0.25%) | Vehicle, Then Reproxalap (0.25%), Then Reproxalap (0.5%) | Total
Number analyzed (Participants) | 22 | 25 | 23 | 70
Age, Customized [Mean (Full Range); unit: years]
  Mean | 45.50 [27 to 66] | 48.84 [28 to 67] | 46.17 [30 to 68] | 46.9 [27 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 14 | 42
  Male | 10 | 9 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 9
  Not Hispanic or Latino | 20 | 23 | 18 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 17 | 13 | 45
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 5 | 14
  Native Hawaiian / Other Pacific Islander | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 5 | 9
  Other - Mixed | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 25 | 23 | 70

OUTCOME MEASURES:

1. Primary Outcome: Subject-Reported Ocular Itching Score
Description: Change from baseline comparison of reproxalap to vehicle for subject-reported ocular itching score from 0 to 212 minutes in the allergen chamber using a 0 -100 millimeter visual analogue scale (0 = none, 100 = severe) was assessed. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included itching score as a dependent variable, treatment, period, and interaction of treatment and period as fixed effects.
Time Frame: Efficacy was assessed from 0 to 212 minutes in the allergen chamber.
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reproxalap (0.25%); Reproxalap (0.5%): Reproxalap was administered once 5 minutes before and 90 minutes after allergen chamber entry.
- Vehicle: Vehicle was administered once 5 minutes before and 90 minutes after allergen chamber entry.
Arm/Group | Reproxalap (0.25%) | Reproxalap (0.5%) | Vehicle
Number analyzed (Participants) | 67 | 69 | 67
units on a scale | 16.410 (1.6195) | 16.964 (1.6150) | 22.310 (1.6188)

2. Secondary Outcome: Subject-Reported Ocular Tearing Score
Description: Change from baseline comparison of reproxalap to vehicle for subject-reported ocular tearing score from 0 to 212 minutes in the allergen chamber using a 4-point scale (0 = none, 3 = severe) was assessed. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included itching score as a dependent variable, treatment, period, and interaction of treatment and period as fixed effects.
Time Frame: Efficacy was assessed from 0 to 212 minutes in the allergen chamber.
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reproxalap (0.25%); Reproxalap (0.5%): Reproxalap was administered twice in a single day.
- Vehicle: Vehicle was administered twice in a single day.
Arm/Group | Reproxalap (0.25%) | Reproxalap (0.5%) | Vehicle
Number analyzed (Participants) | 67 | 69 | 67
units on a scale | 0.8777 (0.0615) | 0.8915 (0.0613) | 1.0507 (0.0614)

3. Secondary Outcome: Investigator-Assessed Conjunctival Redness Score
Description: Change from baseline comparison of reproxalap to vehicle for investigator-assessed conjunctival redness from 0 to 210 minutes in the allergen chamber using a 9-point scale with half unit increments (0 = normal, 4 = prominent) was assessed. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline included itching score as a dependent variable, treatment, period, and interaction of treatment and period as fixed effects.
Time Frame: Efficacy was assessed from 0 to 210 minutes in the allergen chamber.
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reproxalap Ophthalmic Solution (0.5%): Reproxalap was administered twice in a single day.
Arm/Group | Reproxalap (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle
Number analyzed (Participants) | 67 | 69 | 67
units on a scale | 0.5004 (0.0458) | 0.5462 (0.0457) | 0.6497 (0.0458)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately fourteen weeks.
Groups:
- Vehicle Ophthalmic Solution: Vehicle was administered once 5 minutes before and 90 minutes after allergen chamber entry.
Arm/Group | Reproxalap (0.25%) | Reproxalap (0.5%) | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 49/67 | 56/69 | 5/67
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25%) (N=67) | Reproxalap (0.5%) (N=69) | Vehicle Ophthalmic Solution (N=67)
General disorders and administration site conditions (General disorders) | 49 | 56 | 5 — Transient and self-limiting instillation site irritation that resolved in all cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03709121/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT03709121/SAP_001.pdf